CLINICAL TRIAL: NCT00025584
Title: Phase II Trial Of PS-341 In Metastatic Breast Cancer
Brief Title: PS-341 in Treating Women With Metastatic Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02422; ID00-308; N01CM17003 (NIH); CDR0000068976 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-01-23 (Estimated); Status verified 2013-01

CONDITIONS: Recurrent Breast Cancer; Stage IV Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bortezomib

ARMS (1):
- Treatment (bortezomib) (Experimental): Patients receive PS-341 IV over 3-5 seconds twice weekly on weeks 1 and 2. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: bortezomib; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: bortezomib — Given IV
  Other Names: LDP 341; MLN341; VELCADE
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
PS-341 may stop the growth of tumor cells by blocking the enzymes necessary for cancer cell growth. Phase II trial to study the effectiveness of PS-341 in treating women who have metastatic breast cancer

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the efficacy of PS-341, in terms of response rate, in women with metastatic breast cancer.

SECONDARY OBJECTIVES:

I. Determine the clinical activity of this drug, in terms of progression-free survival, in these women.

II. Determine the toxicity profile and tolerability of this drug in these women.

III. Determine the pharmacodynamics of this drug in these women.

OUTLINE:

Patients receive PS-341 IV over 3-5 seconds twice weekly on weeks 1 and 2. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A maximum of 12-35 patients will be accrued for this study within 9-12 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed invasive breast cancer

  * Clinical and/or radiological evidence of stage IV disease
* Relapsed or resistant disease within 6-12 months after completion of prior chemotherapy with doxorubicin or epirubicin and/or paclitaxel or docetaxel foradvanced disease or in the adjuvant setting
* At least 1 unidimensionally measurable lesion

  * At least 20 mm by conventional techniques
  * At least 10 mm by spiral CT scan
  * No bone metastases as only measurable site
  * Pleural or peritoneal effusions not acceptable as measurable disease
* No known brain metastases
* Hormone receptor status:

  * Estrogen receptor-negative
  * Estrogen receptor-positive
* Female
* Performance status - ECOG 0-2
* Performance status - Karnofsky 60-100%
* More than 12 weeks
* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Bilirubin normal
* AST or ALT no greater than 2.5 times upper limit of normal
* Creatinine normal
* Creatinine clearance at least 60 mL/min
* No acute ischemia or significant conduction abnormality by EKG
* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia
* LVEF greater than 50%
* No uncontrolled concurrent illness
* No psychiatric illness or social situation that would preclude study
* No ongoing or active infection
* No prior allergic reaction(s) to compounds of similar chemical or biologic composition to PS-341
* No other malignancy within the past 5 years except carcinoma in situ of the cervix or basal cell skin cancer
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier-method contraception
* See Chemotherapy
* See Disease Characteristics
* No more than 1 prior chemotherapy regimen for metastatic disease

  * High-dose regimen or bone marrow transplantation considered 1 prior regimen
* At least 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin) and recovered
* Prior hormonal therapy for metastatic disease or in adjuvant setting allowed
* Prior localized radiotherapy allowed if it does not influence the signal evaluable lesion
* At least 4 weeks since prior radiotherapy and recovered
* At least 2 weeks since prior minor surgery and recovered
* At least 4 weeks since prior major surgery and recovered
* No other concurrent investigational agent
* No other concurrent investigational or commercial agents or therapies to treat this malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2001-08; Primary Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Objective tumor response (CR + PR) | Up to 24 months
  The agent would be of definite interest for further investigation if the associated response rate is at least 30% (p1), and would not be of further interest if the response rate is below 10% (p0).

SECONDARY OUTCOMES:
Time to progression | Up to 3 years
  Will be reported using the Kaplan-Meier method with 95% confidence intervals indicated.
Overall survival | Up to 3 years
  Will be reported using the Kaplan-Meier method with 95% confidence intervals indicated.
Correlation between variations in the serum levels of adhesion molecules and angiogenic factors | Up to 24 months
  Will be evaluated and descriptive analysis will be performed.
Tissue markers of biological activity | Up to 24 months
  Will be described in case of lesions amenable to tissue biopsy. The plasma pharmacodynamics of PS-341 as measured by the 20S-proteosome assay, will be used to measured the biological activity of the drug and correlated with response to treatment and variations in biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Massimo Cristofanilli, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States